CLINICAL TRIAL: NCT00655083
Title: Pilot Study to Evaluate the Oral Absorption, Safety, and Tolerability of Nepadutant Administered as Single Oral Doses to Infants With Colic and Other Functional Gastrointestinal Disorders
Brief Title: A Phase I Study to Evaluate the Oral Absorption of Nepadutant in Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIC 02; Oral absorption; of Nepadutant in Infants
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Results first posted 2010-08-25 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Infantile Colic; Infantile Functional Gastrointestinal Disorders
Keywords: Infantile colic; Abdominal Cramps; Colicky Pain; Functional gastrointestinal disorders
MeSH Terms: conditions — Colic; Abdominal Pain; Gastrointestinal Diseases | interventions — MEN 11420

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nepadutant 0.1 mg/kg
  Interventions: Drug: Nepadutant
- 2 (Experimental): Nepadutant 0.5 mg/kg
  Interventions: Drug: Nepadutant

INTERVENTIONS:
Drug: Nepadutant — 0.1 mg/Kg as one single oral dose divided in three age strata (from 6 to 24 weeks old)
  Arms: 1
Drug: Nepadutant — 0.5 mg/Kg as one single oral dose divided in three age strata (from 6 to 24 weeks old)
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the gastrointestinal absorption of nepadutant after single dose as oral solution (and the effect of age on its oral absorption) in infants. Oral absorption is evaluated through the drug recovery in urine.

DETAILED DESCRIPTION:
This trial aims to evaluate the oral adsorption of nepadutant (0.1 or 0.5 mg/Kg given as one single dose as oral solution) in infants divided in three age strata (from 6 to 24 weeks old). Oral absorption is evaluated by measuring the amount of nepadutant in the urine output collected during the 24 hours after oral administration with special diapers.

Safety and tolerability of the drug will be evaluated by monitoring any changes in signs/symptoms at medical examination and vital signs during the fist 4 hours post-dose in the Hospital site and then by the parents at home up to 24 hours and 1 week post nepadutant administration.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for inclusion in the study if they meet all of the following criteria:

* Infants with a history consistent with a diagnosis of colic or other functional gastrointestinal disorders
* Age >6 weeks and < 24 weeks
* At least 44 weeks post-conceptual age at enrolment
* Normal growth
* Informed consent by parents (one or both) or legal guardian
* Caregiver available to be trained in collection and storage of used diapers
* Caregiver available to record feeding episodes and defecations on the diary

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

* Clinical evidence of major cardiovascular, respiratory, renal, hepatic, endocrine, metabolic, gastrointestinal (excluding infantile colic and other functional gastrointestinal disorders, unless associated to symptoms which are likely to interfere with drug absorption, e.g. frequent vomiting), haematological, severe dermatological or neurological pathology or other diseases;
* Previous major surgery or blood loss
* Intake of antimuscarinic drugs, simethicone, or dimethicone 24 hours before study treatment administration.

Ages: 6 Weeks to 24 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Blumer, MD, PHD, Study Chair — Rainbow Babies and Children's Hospital
Locations (3):
- United States (3):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kosair Charities Pediatric Clinical Rsearch Unit University of Louisville, Louisville, Kentucky
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period extended from March 2008 to May 2009 at three Hospital Clinics
Pre-assignment Details: Twenty out of the 21 enrolled infants were treated with study medication (1 infant did not attend the clinic after screening). NOTE: although the goal was to enroll 24 subjects, slow subject enrollment and expired drug restricted enrollment to 20 subjects
Groups:
- Nepadutant 0.1 mg/kg: Nepadutant 0.1 mg/kg
- Nepadutant 0.5 mg/kg: Nepadutant 0.5 mg/kg
Period: Overall Study
Arm/Group | Nepadutant 0.1 mg/kg | Nepadutant 0.5 mg/kg
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepadutant 0.1 mg/kg | Nepadutant 0.5 mg/kg | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Customized [Number; unit: participants]
  Age Group 6 to <12 weeks | 4 | 3 | 7
  Age Group 12 to <18 weeks | 4 | 5 | 9
  Age Group 18 to 24 weeks | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Drug Concentration Measurement in the Urine Collected by Diapers Along 24 Hours Post Dose and One Week After Dose in All Treated Infants and by Age and Dose Subgroups.
Description: Nepadutant was measured in the 24-h urine collection post both doses (0.1 and 0.5 mg/kg dose), in the age strata 6-<12 and 12-<18 weeks, using urinary collection/extraction from pre-weighed special fiber based diapers.
Time Frame: 24 hours
Population: Urinary drug concentration was analysed by dose and age stratum of the infants (6-<12 and 12- <18 weeks of age). Imputation technique was adopted for urine samples highly contaminated by faeces.
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Nepadutant 0.1 mg/kg | Nepadutant 0.5 mg/kg
Number analyzed (Participants) | 8 | 8
ng
  6- <12 week old | 5041 (7081) | 6474 (2463)
  12- < 18 week old | 2095 (1151) | 3727 (2845)

2. Secondary Outcome: Number of Adverse Events After Administration of Single Oral Doses up to 0.5 mg/kg of Nepadutant in Infants.
Description: Number of adverse events (AE) reported by dose and age stratum 6-<12 and 12-<18 weeks.
Time Frame: one week
Population: Number of adverse events by dose and age strata (6-<12 and 12- <18 weeks of age) are reported by system organ class and preferred term.
Measure: Number; unit: Adverse Events
Arm/Group | Nepadutant 0.1 mg/kg | Nepadutant 0.5 mg/kg
Number analyzed (Participants) | 8 | 8
Adverse Events
  6- <12 week old | 0 | 3
  12- < 18 week old | 1 | 1

3. Primary Outcome: Drug Concentration Measurement in the Urine Collected by Diapers Along 24 Hours Post Dose and One Week After Dose in All Treated Infants and by Age and Dose Subgroups.
Description: Nepadutant was measured in the 24-h urine collection post both doses (0.1 and 0.5 mg/kg dose), in the age stratum 18-24 weeks, using urinary collection/extraction from pre-weighed special fiber based diapers.
Time Frame: 24 hours
Population: Urinary drug concentration was analysed by dose and age stratum of the infants (18-24 weeks of age). Imputation technique was adopted for urine samples highly contaminated by faeces.
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Nepadutant 0.1 mg/kg | Nepadutant 0.5 mg/kg
Number analyzed (Participants) | 4 | 0
ng | 1127 (1032) |

4. Secondary Outcome: Number of Adverse Events After Administration of Single Oral Doses up to 0.5 mg/kg of Nepadutant in Infants.
Description: Number of adverse events (AE) reported by dose and age stratum 18-24 weeks.
Time Frame: one week
Population: Number of adverse events by dose and age stratum (18-24 weeks of age) are reported by system organ class and preferred term.
Measure: Number; unit: Adverse Events
Arm/Group | Nepadutant 0.1 mg/kg | Nepadutant 0.5 mg/kg
Number analyzed (Participants) | 4 | 0
Adverse Events | 3 |

ADVERSE EVENTS:
Time Frame: Adverse events were recorded after 24 hours after dosing and at 1 week final follow up.
Arm/Group | Nepadutant 0.1 mg/kg | Nepadutant 0.5 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 4/12 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nepadutant 0.1 mg/kg (N=12) | Nepadutant 0.5 mg/kg (N=8)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) — mild, possibly tretment related, 2 days after dosing lasting < 1 day
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — mild, unlikely treatment related
hard stools (Gastrointestinal disorders) | 1 (1) | 0 (0) — mild, possibly treatment related, 2 hours post dosing and lasting up to the following day
pyrexia (General disorders) | 1 (1) | 1 (1) — mild, unlikely treatment related
dermatitis by diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — mild, unlikely treatment related
middle ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) — mild, unlikely treatment related
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — mild, unlikely treatment related

LIMITATIONS AND CAVEATS:
No infants aged 18-24 weeks were dosed at 0.5 mg/kg dose when the trial was stopped because of slow recruitment and drug expiration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less